CLINICAL TRIAL: NCT01875770
Title: Continuing Assessment of Patients Treated With ranibizUmab for REtinal Vein Occlusion (CAPTURE)
Acronym: CAPTURE
Status: Terminated | Type: Observational
Why Stopped: The study was terminated as patients could not be followed-up during the COVID pandemic. Since this was a non-intervention study, as per Johns Hopkins University policy, we had to hold off the patient visits during the pandemic.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: NA_00079952
Record Dates: First submitted 2013-06-10; First posted 2013-06-12 (Estimated); Last update posted 2021-10-12 (Actual); Status verified 2021-05

CONDITIONS: Retinal Vein Occlusion
Keywords: Retinal Vein Occlusion
MeSH Terms: conditions — Retinal Vein Occlusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Treated with Ranibizumab in previous trial: Treated with Ranibizumab in previous trial

SUMMARY:
This research is being done to assess the long term prognosis of patients treated with ranibizumab for edema due to retinal vein occlusion.

DETAILED DESCRIPTION:
People treated with ranibizumab for edema due to retinal vein occlusion as part of previous studies at the Wilmer Eye Institute and who are currently being seen by their ophthalmologist at the Wilmer Eye Institute are followed up to assess long term outcomes

ELIGIBILITY:
Inclusion Criteria:

* All patients who have been enrolled in the following three trials will be included in the study:

A) "A Pilot, Open-Label Study of the Safety, Tolerability, and Bioactivity of Multiple Intravitreal Injections of Ranibizumab in Subjects with Macular Edema Secondary to Vein Occlusions.", B) "Extended follow-up of patients with macular edema due to bRanch rETinal vein occlusion (BRVO) or centrAl retinal veIn occlusioN (CRVO) previously treated with intravitreal ranibizumab (RETAIN) " C) "RanibizumabDosE Comparison (0.5mg and 2.0mg) and the Role of LAser in the ManagemenT of REtinal Vein Occlusion - A Pharmacodynamic Approach (RELATE)"

Exclusion Criteria:

* None

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who have been enrolled in the following three trials will be included in the study:
  A) "A Pilot, Open-Label Study of the Safety, Tolerability, and Bioactivity of Multiple Intravitreal Injections of Ranibizumab in Subjects with Macular Edema Secondary to Vein Occlusions.", B) "Extended follow-up of patients with macular edema due to bRanch rETinal vein occlusion (BRVO) or centrAl retinal veIn occlusioN (CRVO) previously treated with intravitreal ranibizumab (RETAIN) " C) "RanibizumabDosE Comparison (0.5mg and 2.0mg) and the Role of LAser in the ManagemenT of REtinal Vein Occlusion - A Pharmacodynamic Approach (RELATE)"
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2018-10-11 (Actual); Study Completion 2021-03-03 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in BCVA at 5 and 10 years. | 10 years
  Mean change from baseline in BCVA at 5 and 10 years.

SECONDARY OUTCOMES:
Mean change from baseline in foveal thickness at 5 and 10 years | 10 years
  Mean change from baseline in foveal thickness at 5 and 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter Campochiaro, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Wilmer Eye Institute, Baltimore, Maryland, United States